CLINICAL TRIAL: NCT01234519
Title: A Phase I/II Trial of AEZS-108 in Locally Advanced Unresectable or Metastatic Luteinizing Hormone-releasing Hormone(LHRH) Positive Urothelial Carcinoma Patients Who Failed Platinum Based Chemotherapy
Brief Title: A Phase I/II Trial of AEZS-108 in Urothelial Cancer Patients Who Failed Platinum-chemotherapy
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Poor recruitment
Sponsor: AEterna Zentaris (Industry)
Collaborators: University of Miami (Other); Miami VA Healthcare System (U.S. Federal Agency); University of Miami Sylvester Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AEZS-108-046; EProst # 20091095 (Other: Sylvester Comprehensive Cancer Center)
Record Dates: First submitted 2010-11-02; First posted 2010-11-04 (Estimated); Last update posted 2018-03-15 (Actual); Status verified 2013-03

CONDITIONS: Urothelial Carcinoma
Keywords: ureter cancer; renal pelvis cancer; bladder cancer; urethra
MeSH Terms: conditions — Carcinoma, Transitional Cell; Ureteral Neoplasms; Urinary Bladder Neoplasms | interventions — LHRH, lysine(6)-doxorubicin

STUDY DESIGN:
Intervention Model Description: Phase 1 : conventional 3+3 design. Phase 2: Simon's two-stage design will be utilized. In Stage I, 22 patients will be treated with the dose determined in Phase I. The study will be terminated for futility if no more than 2 patients out of the 22 patients in Stage I are responders. If 3 or more responders are observed, an additional 18 patients will be enrolled. If at least 8 out of the 40 patients are responders, the treatment will be considered worthy of further development.
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Phase 1 - Cohort 1 (Experimental): Determination of maximum tolerated dose (MTD) and recommended parenteral administration dosing for AEZS-108 in 4 sequential cohorts of patients (3-6 patients/cohort).
  Patients will be enrolled in cohorts of 3 at a specified AEZS-108 dose beginning with 160mg/m^2. Enrollment will be suspended until all members of a cohort have been observed for dose limiting toxicities (DLT) for a period of 3 weeks (1 cycle of AEZS-108) from initial treatment with AEZS-108. Dose escalation will proceed within each cohort according to a specific scheme where DLT is defined.
  Interventions: Drug: AEZS-108
- Phase 1 - Cohort 2 (Experimental): Determination of maximum tolerated dose (MTD) and recommended parenteral administration dosing for AEZS-108 in 4 sequential cohorts of patients (3-6 patients/cohort).
  Interventions: Drug: AEZS-108 at MTD
- Phase 1 - Cohort 3 (Experimental): Determination of maximum tolerated dose (MTD) and recommended parenteral administration dosing for AEZS-108 in 4 sequential cohorts of patients (3-6 patients/cohort).
  Interventions: Drug: AEZS-108
- Phase 1 - Cohort 4 (Experimental): Determination of maximum tolerated dose (MTD) and recommended parenteral administration dosing for AEZS-108 in 4 sequential cohorts of patients (3-6 patients/cohort).
  Interventions: Drug: AEZS-108
- Phase 2 (Experimental): AEZS-108 at MTD to determine efficacy in up to 40 patients.
  Interventions: Drug: AEZS-108

INTERVENTIONS:
Drug: AEZS-108 — 128, 160, 210 or 267 mg/m2, 2-hour intravenous (IV) infusion, Day 1 of 21-day cycles , until toxicity or progression, up to 6 cycles
  Other Names: ZEN-008; AN-152; D-81858
  Arms: Phase 1 - Cohort 1; Phase 1 - Cohort 3; Phase 1 - Cohort 4; Phase 2
Drug: AEZS-108 at MTD — 2-hour IV infusion, Day 1 of 21-day cycles , until toxicity or progression, up to 6 cycles
  Other Names: ZEN-008; AN-152; D-81858
  Arms: Phase 1 - Cohort 2

SUMMARY:
The purpose of this study is to determine the appropriate dose of AEZS-108 to treat patients with a tumor of the urinary system.

DETAILED DESCRIPTION:
AEZS-108 is an investigational drug, combining luteinizing hormone-releasing hormone (LHRH), an hormone and doxorubicin (a drug approved to treat different types of cancer).

Some tumors, such as those found in the urinary system (also called urothelial carcinomas), have LHRH hormone receptors to which the LHRH hormone part of AEZS-108 is attracted.

AEZS-108 is expected to work by accumulating mostly on the surface of cancer cells that have LHRH hormone receptors and by delivering doxorubicin more directly into the cells to kill them. This would allow the use doxorubicin at lower doses and thus would cause less toxicity.

In the first part of the study, the appropriate dose of AEZS-108 will be determined based on its side effects. The best dose will be the highest one without severe side effects.

In the second part of the study, this best dose of AEZS-108 will be given to determine its efficacy to stop the tumor from progressing.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed locally advanced or metastatic urothelial carcinoma
* Expression of LHRH receptors confirmed by immunohistochemistry on archival cancer tissue
* Measurable disease on radiological studies
* Patients with Locally advanced unresectable or metastatic urothelial carcinoma
* Documented progression on at least one prior chemotherapy regimen which must have incorporated platinum based therapy
* Left ventricular ejection fraction (EF) > 50%
* Eastern cooperative oncology group (ECOG) status of 0, 1 or 2
* Adequate bone marrow, renal and hepatic function

Exclusion Criteria:

* Prior treatment with or allergy to any components of AEZS-108
* Active second malignancies other than non-melanoma skin cancers
* Ongoing use of an LHRH agonist (or antagonist)
* Presence of an active infection or fever > 38.5 C, parenchymal brain metastases or uncontrolled intercurrent illness
* Prior exposure to anthracyclines or anthracenediones including doxorubicin, daunorubicin, and mitoxantrone
* Patients who received radiotherapy within 4 weeks of entry
* Major surgery within the last 4 weeks and minor surgery in last 7 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-11; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | Day 1 of each 21-day cycle
  Toxicity per Common Terminology Criteria for Adverse Events (CTCAE).

SECONDARY OUTCOMES:
Objective tumor response | Within 5 days of cycle 4, then every 3 cycles
  Response evaluation criteria in solid tumors (RECIST) criteria.
Progression-free survival (PFS) | last cycle
  Time elapsed from the start of treatment to the date of documented progression or death, whichever comes first.
Pharmacokinetics (PK) | cycle 1
  To evaluate PK parameters of a single dose AEZS-108 and explore whether the PK parameters are associated with cardiac effects as measured by electrocardiography.
Overall survival | last cycle
  Time elapsed from the start of treatment until death.
Circulating tumor cell (CTC) levels | last cycle
  To quantify tumor cells and attempt to correlate their presence and response to the outcomes of this study.

CONTACTS AND LOCATIONS:
Overall Officials: Gustavo Fernandez, MD, Principal Investigator — University of Miami
Locations (2):
- United States (2):
  - University of Miami Miller School of Medicine, Miami, Florida
  - Univerity of Pennsylvania, Philadelphia, Pennsylvania